CLINICAL TRIAL: NCT02828410
Title: Evaluating the Nutritional Impact of Serum-Derived Bovine Immunoglobulin Protein Isolate in Subjects With Ileal Pouch-Anal Anastomosis
Brief Title: Nutritional Impact of Serum-Derived Bovine Immunoglobulin Protein Isolate in Subjects With IPAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Entera Health, Inc (Industry)
Responsible Party: Principal Investigator, Francis Farraye, MD, BMC Investigator, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33890
Record Dates: First submitted 2016-07-02; First posted 2016-07-11 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pouchitis; Irritable Pouch Syndrome
Keywords: serum bovine immunoglobulin protein isolate; IPAA; quality of life
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBI (Experimental): Serum bovine immunoglobulin protein isolate (SBI)
  Interventions: Dietary Supplement: SBI

INTERVENTIONS:
Dietary Supplement: SBI — Serum bovine immunoglobulin protein isolate 10 g twice per day
  Other Names: EnteraGam

SUMMARY:
This is an open label trial to test the hypothesize that serum bovine immunoglobulin protein isolate (SBI) will improve the nutritional status and quality of life (QOL) of patients with an ileal pouch anal anastomosis (IPAA) and symptoms of pouchitis. Subjects with symptomatic IPAA will receive two packets of EnteraGam twice daily (total daily dose of 20 g SBI) for up to 24 weeks. The primary objective of this study is to determine whether SBI therapy leads to improved nutritional status and QOL. A secondary objective is to evaluate SBI in the management of their disease, including impact on clinical symptoms.

DETAILED DESCRIPTION:
This is an open-label study involving patients who are status post ileal pouch-anal anastomosis age 18 and 75 who receive care at Boston Medical Center's Center for Digestive Disorders (CDD). There is no randomization or use of placebo in this study and patients will be recruited sequentially. This is an open-label, single center study evaluating the effectiveness of SBI or EnteraGam (10.0 g twice per day) on nutritional status and quality of life in patients with ileal pouch-anal anastomosis.

Nutritional status and inflammation be assessed by measuring CBC with differential, vitamin D, vitamin B12, pre-albumin, albumin, ferritin, ESR, CRP, alpha-1-antitrypsin, and fecal calprotectin levels at screening, Day 84, and Day 168. Stool samples from these same time points will also be frozen and stored until the end of the study for potential fecal microbiome analysis depending on the results of other outcome measures.

The effect of SBI on a subject's quality of life (QoL) will be evaluated using the Short Inflammatory Bowel Disease Questionnaire and Cleveland Global Quality of Life scores at baseline, Day 28, Day 84, and End of Study.

The short form of disease specific QoL (s-IBDQ) includes 10 questions derived from the 32 questions IBDQ concerning QoL. It covers four items: bowel symptoms, systemic symptoms, emotional, and social functions. The total score ranges from 10 (worst health) to 70 (best health).

The Cleveland Global Quality of Life (CGOL) score is an instrument specifically designed for patients with ileal pouches. Subjects will be asked to rate each of three items (current QOL, current quality of health, and current energy level) on a scale of 0-10, 0 being the worst and 10 the best. The sum of the three scores divided by 30 will provide the CGQL score.

The Modified Pouchitis Disease Activity Index (mPDAI) will be used to evaluate for pouchitis and assess the overall disease activity for each subject at baseline pouchoscopy. This modified diagnostic instrument consists of two component scores: clinical symptoms (range 0-6 points) and endoscopic appearence (range 0-6 points). Follow-up pouchoscopy is not part of the study protocol. However, if a patient warrants follow-up pouchoscopy at any point during the study period based on standard of care (most likley due to worsening or non-responsive symptoms), then the mPDAI at follow-up pouchoscopy will also be calculated and included in outcomes analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between the ages of 18-75 years, inclusive.
* Patient has history of UC or Crohn's disease (CD) diagnosed by standard clinical, radiographic, endoscopic, and histopathological criteria.
* Patient has undergone total proctocolectomy and IPAA surgery a minimum of 6 months prior to screening.
* Patient has symptoms suggestive of pouchitis including frequent bowel movements of greater than or equal to seven per day (≥7 per day), and one or more of the following: daily rectal bleeding, fecal urgency, abdominal cramps, or fever >37.8oC).
* Patient is capable of understanding the requirements of the study and has signed / dated an IRB approved informed consent form.

Exclusion Criteria:

* Patient cannot or will not provide written informed consent.
* Patient has a known allergy or hypersensitivity to beef, beef products, or any ingredient used in EnteraGam.
* Patient has clinical signs and symptoms of an active infection.
* Patient is on antibiotic therapy (other than for pouchitis treatment) at any time in the 30 days prior to screening.
* Patient has active alcohol or drug abuse or psychiatric disorders felt to preclude his / her ability to complete the study.
* Patient who, in the opinion of the investigator, has a poorly controlled / uncontrolled significant medical condition that would interfere with the study.
* Positive stool test (PCR) for C. difficile.
* Use of antidiarrheal medications (ADM). - Exception: patients who, in the opinion of the Investigator, are on stable treatment with ADMs may be enrolled provided that the administration schedule is intended to be maintained or decreased during the study and the subject has been on stable treatment with ADMs for at least 30 days prior to screening; otherwise, these agents are prohibited in the study.
* Use of an investigational product or participation in a clinical trial within the past three months.
* Use of a biologic (e.g., infliximab, adalimumab) within the last 3 months.
* Patient is pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
BMI | 6 months
Pre-albumin | 6 months
Albumin | 6 months
Vitamin D | 6 months
Vitamin B12 | 6 months
Ferritin | 6 months
Short Inflammatory Bowel Disease Quality of Life Score | 6 months
Cleveland Global Quality of Life Score | 6 months

SECONDARY OUTCOMES:
Nocturnal Bowel Movements | 6 months
  Average number of nightly nocturnal bowel movements over the past week
Concomitant Medications | 6 months
Abdominal Cramping | 6 months
  Number of days experiencing abdominal cramping over the past week
Consistency of Bowel Movements | 6 months
  Average Bristol Stool Scale score for bowel movements during the previous week
Incontinence | 6 Months
  Number of incontinence episodes over the past week
ESR | 6 Months
  Sedimentation Rate
CRP | 6 Months
  C-reactive protein
Fecal calprotectin | 6 Months
Alpha-1-antitrypsin | 6 Months
Number of Bowel Movements | 6 Months
  Average number of daily bowel movements over the past week
Fecal Urgency | 6 Months
  Average number of days with fecal urgency over the past week
Modified Pouchitis Disease Activity Index Score | 6 Months
  When applicable
Rectal Bleeding | 6 Months
  Average number of days with rectal bleeding over the past week

CONTACTS AND LOCATIONS:
Overall Officials: Francis Farraye, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No